CLINICAL TRIAL: NCT02044588
Title: The Outcomes of Kidney Transplantation Between Recipients Receiving Graft From Donors With Positive and Negative HBsAg
Brief Title: Hepatitis B Antigen Kidney Graft Into Protective Level Hepatitis B Antibody Recipients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Wiwat Chancharoenthana, Division of Nephrology, Department of Medicine, Faculty of Medicine, Chulalongkorn University
Other Study IDs: WWC-001
Record Dates: First submitted 2014-01-20; First posted 2014-01-24 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: HBsAg(+) Donor Kidney Allograft; HBsAg(-) Donor Kidney Allograft
Keywords: HBsAg(+) donor; HBsAg(-) donor; Anti-hepatitis B antibody; Kidney allograft
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HBsAg negative kidney allograft donor
- HBsAg positive kidney allograft donor: HBsAg positive kidney allograft donor
  Interventions: Biological: HBsAg positive kidney allograft donor

INTERVENTIONS:
Biological: HBsAg positive kidney allograft donor
  Groups: HBsAg positive kidney allograft donor

SUMMARY:
To determine the safety of using kidney organ from hepatitis B surface antigen positive donor, the author conducted the single-center, prospective study of the use of these kidneys for recipients who have protective level of hepatitis B surface antibodies.

DETAILED DESCRIPTION:
The kidney transplant registry was conducted in KCMH since the year of 2000 until the present.

The inclusion criterion was:

* All kidney allograft recipients who received at least one month after transplantation.
* All kidney recipients who already had the protective antibody against hepatitis B virus infection defined by anti-HBs titer above 100 mIU/mL at pre-transplantation period.

The exclusion criterion was:

* The recipients with positive hepatitis C virus antibody.
* The recipients who had received a previous or simultaneous non-kidney solid organ transplant.
* The recipients those lost to follow-up.

Study group:

* The recipients who received kidney allograft from the HBsAg(+) donor.

Control group:

* The recipients who received kidney allograft from the HBsAg(-) donor.

According to the Thai Red Cross National Organ Donation and our institute's policy, the HBsAg(+) kidney allografts were distributed to only and informed consent.

Data collection:

* Baseline characteristic data e.g. donor and recipient age, donor and recipient gender, HLA, PRA, anti-HBs titer, immunity against HBV status (both natural and vaccinated),immunosuppressive regimens were collected.
* The recipients were prospective followed up at month 3, 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, 120.
* Clinical data including jaundice, hepatitis, graft rejection were collected
* Laboratory data of HBsAg, anti-HBc, HBV DNA, SGOT, SGOT, eGFR were collected.
* Pathological data of allograft biopsy at month 12 and 24 were retrieved.

Outcomes:

* Primary outcome: hepatitis B transmission rate.
* Secondary outcome: graft survival, patient survival.

ELIGIBILITY:
The inclusion criterion was:

* All kidney allograft recipients who received at least one month after transplantation.
* All kidney recipients who already had the protective antibody against hepatitis B virus infection defined by anti-HBs titer above 100 mIU/mL at pre-transplantation period.

The exclusion criterion was:

* The recipients with positive hepatitis C virus antibody.
* The recipients who had received a previous or simultaneous non-kidney solid organ transplant.
* The recipients those lost to follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All kidney transplant recipients from January 1, 2000 until the present (upto year 2013) were prospective follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2000-01; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Hepatitis B transmission rate | January 2000 to December 2013
  The hepatitis B transmission rate was determined at month 3, 6, 9, 12, 18, 24, 36, 48, 60, 72, 84, 96, 108, 120 by using:
  * Clinical data including jaundice, hepatitis, acute liver failure.
  * Laboratory data of HBsAg, anti-HBc, HBV DNA, SGOT, SGOT.
  * Radiological data of liver ultrasonography.

SECONDARY OUTCOMES:
Graft survival rate | January 2000 to December 2013
  The graft survival rate was determined by Kaplan-Meyer survival analysis.

OTHER OUTCOMES:
Patient survival rate | January 2000 to December 2013
  The patient survival rate was determined by Kaplan-Meyer survival analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Wiwat Chancharoenthana, MD, MSc, Principal Investigator — Chulalongkorn University
Locations (1):
- Wiwat Chancharoenthana, Bangkok, Bangkok, Thailand

REFERENCES:
- [Derived] Chancharoenthana W, Townamchai N, Pongpirul K, Kittiskulnam P, Leelahavanichkul A, Avihingsanon Y, Suankratay C, Wattanatorn S, Kittikowit W, Praditpornsilpa K, Tungsanga K, Eiam-Ong S. The outcomes of kidney transplantation in hepatitis B surface antigen (HBsAg)-negative recipients receiving graft from HBsAg-positive donors: a retrospective, propensity score-matched study. Am J Transplant. 2014 Dec;14(12):2814-20. doi: 10.1111/ajt.12921. Epub 2014 Nov 13. PMID 25395260